CLINICAL TRIAL: NCT03051932
Title: Effects of Intravenous Acetaminophen in Patients Undergoing Thoracoscopic Surgery
Acronym: IVTylenol
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Not funded
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-0340
Record Dates: First submitted 2017-01-30; First posted 2017-02-14 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2017-12

CONDITIONS: Post-thoracotomy Pain Syndrome
MeSH Terms: interventions — Acetaminophen; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ofiramev®( IV Acetaminophen) (Active Comparator): Patients randomized to the treatment arm will receive 1 g (100 mL) intravenous acetaminophen infused over 15-minutes every 6 hours for 4 doses total.
  Interventions: Drug: Ofiramev® (IV Acetaminophen)
- Placebo IV administration (Placebo Comparator): Patients randomized to the placebo arm will receive 100 mL of normal saline infused over 15 minutes every 6 hours for 4 doses total
  Interventions: Drug: Placebo IV administration

INTERVENTIONS:
Drug: Ofiramev® (IV Acetaminophen) — Post -op pain medication
  Other Names: IV Tylenol
  Arms: Ofiramev®( IV Acetaminophen)
Drug: Placebo IV administration — Post -op pain
  Other Names: Normal Saline
  Arms: Placebo IV administration

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled trial. A total of 100 patients, 50 per treatment arm, undergoing minimally invasive thoracic surgery will be randomized 1:1 across 2 treatment arms: Ofiramev® (acetaminophen) injection 1,000 mg (100 mL) plus patient-controlled analgesia (PCA) and 100 mL placebo plus PCA.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, placebo-controlled trial. A total of 100 patients, 50 patient per treatment arm, undergoing minimally invasive thoracic surgery will be randomized 1:1 across 2 treatment arms: Ofiramev® (acetaminophen) injection 1,000 mg (100 mL) plus patient-controlled analgesia (PCA) and 100 mL placebo plus PCA. All patients will be enrolled from a single site.50 patient will be enrolled in each arm (placebo/ acetamophin). Each subject will be administered a single dose of study drug or placebo infused over 15-minutes, four times, six hours apart. The duration of subject participation will be ten weeks. Total duration of the study is expected to be 52 weeks. The primary endpoints of the study will be the amount of postoperative narcotic used, patient assessment of pain as measured by a validated pain survey, and length of stay in the hospital.

For postoperative pain assessment, the Numeric Rating Scale (NRS) will be used (NRS: 0-10; 0: no pain, 10: worst pain imaginable). Pain will be evaluated at 2-hour intervals in the post-anesthesia care unit followed by 4-hour intervals once the patient is transferred to the floor. Nurses who are blinded to the analgesic method will evaluate pain levels. Hospital length of stay will be measured from date of admission to date of discharge.

The study drug, Ofiramev® (acetaminophen) injection is a non-salicylate antipyretic and non-opioid analgesic agent. The precise mechanism of the analgesic and antipyretic properties of acetaminophen is not established but is thought to primarily involve central actions. The study drug is a clear, colorless formulation of acetaminophen intended for intravenous infusion and is packaged in glass vials containing 100 mL of 1000 mg acetaminophen (10 mg/mL). The investigational pharmacy will transfer the study drug to a 100 mL bag. The placebo solution will consist of 100 mL normal saline in an identical 100 mL bag with identical labeling. Prior to the induction of anesthesia subjects will receive a single dose of Ofiramev® or placebo by IV infusion over 15 minutes. Following the first dose, each subsequent dose will be given every 6 hours for a total of 4 doses. Regardless of treatment arm, study drug and placebo will be dispensed in the same manner.

Investigational drugs are stored in the investigational drug service storeroom and/or pharmacy satellite depending on the nature of the drug study. All study drug inventory is labeled with IRB identification and stored separately from other commercial drug products under appropriate security and stability conditions. OFIRMEV should be stored at 20°C to 25°C (68°F to 77°F) and should be used within 6 hours after opening.

An accurate and current accounting of the dispensing and return of study drug for each subject will be maintained on an ongoing basis by a member of the study site staff. The number of study drug dispensed and returned by the subject will be recorded on the Investigational Drug Accountability Record. The study monitor will verify these documents throughout the course of the study.

Patients can voluntarily withdraw from the trial for any reason at any time. Subjects will be withdrawn from the study in the event of unplanned conversion to open thoracic surgery or administration of neuraxial opioids. If a subject is withdrawn from treatment due to an adverse event, the subject will be followed and treated by the Investigator until the abnormal parameter or symptom has resolved or stabilized.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-99 years
* Undergo minimally invasive thoracic surgery at UTMB
* Weight > 50 kg
* Written informed consent obtained from subject

Exclusion Criteria:

* Hepatic dysfunction
* Renal dysfunction
* Chronic alcohol consumption
* Acetaminophen sensitivity
* Opioid tolerance
* History of chronic pain
* Vulnerable populations including pregnant and prisoners
* Extension into an extrathoracic compartment (i.e. minimally invasive esophagectomy), or concomitant chest wall resection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
The amount of postoperative narcotic used. | Within 7 days of surgery
  the amount of postoperative narcotic used, after surgery.

SECONDARY OUTCOMES:
The amount of postoperative pain. | An average of 4 days
  The amount of postoperative patient assessment of pain as measured by a validated pain survey (NRS)
length of stay in the hospital | An average of 4 days
  length of stay in the hospital from admission to discharge of patient after surgery.
The amount of postoperative pain. | Within 2-4 weeks of surgery
  The amount of postoperative patient assessment of pain as measured by patient satisfaction survey on 2-4 weeks post-op clinic follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ikenna Okereke, MD, Principal Investigator — The University of Texas Medical Branch, Galveston

IPD SHARING:
Plan to Share IPD: Undecided